CLINICAL TRIAL: NCT05000112
Title: The Influence of Vaginal Microbiome-host Interaction in the Mechanism of Mesh Exposure After Trans-Vaginal Mesh Implantation
Brief Title: Vaginal Microbiome-host Interaction in Mesh Exposure After TVM Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-2936
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-07

CONDITIONS: Vaginal Microbiome; Graft Versus Host Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with mesh exposure: During the physical examination, a speculum was inserted into the vagina to observe the vaginal epithelium for mesh exposure. If the mesh is seen on surface of the vaginal mucosa, the patient is diagnosed with mesh exposure.
- Patients without mesh exposure: During the physical examination, a speculum was inserted into the vagina to observe the vaginal epithelium for mesh exposure. If the mesh is not seen on surface of the vaginal mucosa, bimanual examination will be performed to confirm no foreign body can be feeled on surface of the vaginal mucosa. Then the patient belong to this group.

SUMMARY:
Transvaginal pelvic mesh implantation（TVM） is a foreign body implantation operation with intraoperative colonization of vaginal bacteria. However, the vaginal microbiome-host interaction and its influence in the mechanism of mesh exposure after TVM remains unclear. This study will enroll post-TVM patients with and without mesh exposure and use their vaginal swabs to perform TRACE-seq and cytokine analysis. The microbiome-host interactions related with mesh exposure and the changes in protein expression will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with "III-IV degree uterine/apex/anterior vaginal wall prolapse and I-II degree of posterior vaginal wall prolapse" who agree to be treated by transvaginal pelvic mesh implantation.
* All surgeries were performed by surgeons with extensive experience in transvaginal mesh implantation (>20 vaginal mesh implantation per year) using macroporous, monofilament, polypropylene mesh.

Exclusion Criteria:

* 1. Have had sex in the past 5 days or had vaginal irrigation;
* 2. Use oral or vaginal antibiotics, antifungal, immunosuppressant, hormone drugs or probiotics for the last 30 days.
* 3. Combined with immunosuppressive diseases, diseases with contraindication of vaginal estrogen such as breast cancer, endometrial cancer.
* 4. If the patient has a uterus before surgery and does not undergo total transvaginal hysterectomy during surgery,
* 5. Intraoperative bladder injury or intraoperative hemorrhage >500ml or postoperative hematoma.

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with "III-IV degree uterine/apex/anterior vaginal wall prolapse and I-II degree of posterior vaginal wall prolapse" who agree to be treated by transvaginal pelvic mesh implantation. All surgeries were performed by surgeons with extensive experience in transvaginal mesh implantation (>20 vaginal mesh implantation per year) using macroporous, monofilament, polypropylene mesh.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiome-host interaction in patients after TVM | Over 6 months postoperative
Vaginal microbiome-host Interaction associated with mesh exposure after TVM | Over 6 months postoperative

SECONDARY OUTCOMES:
Difference of vaginal microbiome between groups | Over 6 months postoperative
Differentially expressed genes in host-mesh interaction between groups | Over 6 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College